CLINICAL TRIAL: NCT07244939
Title: Cephea South America Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10554
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-11

CONDITIONS: Mitral Regurgitation; Mitral Stenosis
Keywords: Symptomatic mitral valve disease; Cephea Mitral Valve System
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Cephea TMVR (Experimental): Treatment of symptomatic patients with mitral valve disease (including mitral regurgitation, mitral stenosis and mixed mitral valve disease) with the Cephea Mitral Valve System
  Interventions: Device: Cephea Mitral Valve System

INTERVENTIONS:
Device: Cephea Mitral Valve System — Cephea Mitral Valve System

SUMMARY:
The objective of this study is to evaluate the preliminary safety and effectiveness of the Cephea Mitral Valve System for the treatment of symptomatic patients with mitral valve disease (including mitral regurgitation, mitral stenosis and mixed mitral valve disease) in whom transcatheter therapy is deemed more appropriate than open heart surgery.

ELIGIBILITY:
Key Inclusion Criteria:

* Mitral valve disease resulting in mitral regurgitation (MR ≥ Grade III) and/or severe mitral valve stenosis (mitral valve area ≤ 1.5cm²) per American Society of Echocardiography criteria
* LVEF ≥ 30%
* In the judgement of the Site Heart Team, transcatheter therapy is deemed more appropriate than open heart surgery

Key Exclusion Criteria:

* Prior surgical or interventional treatment that interferes with the Cephea valve delivery or function
* Need for emergent or urgent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Freedom from all-cause mortality | 30 days post implant
  Primary Safety Endpoint
Reduction of MR to ≤ Grade I | 30 days post implant
  Primary Effectiveness Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Barathi Sethuraman, Study Director — Abbott Structural Heart
Locations (3):
- Instituto do Coracao (InCor) - HCFMUSP, São Paulo, Brazil
- Chile (2):
  - Instituto Nacional del Torax, Santiago
  - Hospital Clinico San Borja Arriarán, Santiago